CLINICAL TRIAL: NCT04224532
Title: The Effect of Pneumoperitoneum Timing on Intracranial Pressure in Laparoscopic Cholecystectomy: Before or After Reverse Trendelenburg Position
Brief Title: The Effect of Pneumoperitoneum Timing on Intracranial Pressure in Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019.10.103.072
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-01

CONDITIONS: Intracranial Pressure Increase; Pneumoperitoneum
Keywords: optic nerve sheath diameter; intracranial pressure; laparoscopic cholecystectomy; pneumoperitoneum
MeSH Terms: conditions — Intracranial Hypertension; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Pneumoperitoneum is induced before reverse Trendelenburg position.
  Interventions: Procedure: Pneumoperitoneum Timing (Before Positioning)
- Group RT (Experimental): Pneumoperitoneum is induced after reverse Trendelenburg position.
  Interventions: Procedure: Pneumoperitoneum Timing (After Positioning)

INTERVENTIONS:
Procedure: Pneumoperitoneum Timing (Before Positioning) — Before Reverse Trendelenburg Position
  Arms: Group P
Procedure: Pneumoperitoneum Timing (After Positioning) — After Reverse Trendelenburg Position
  Arms: Group RT

SUMMARY:
Reverse Trendelenburg position has been shown to slightly reduce the intracranial pressure associated with pneumoperitoneum. However, there are no studies on the effect of the timing of reverse Trendelenburg position on intracranial pressure. This study will monitor the effect of reverse Trendelenburg position before or after pneumoperitoneum on intracranial pressure and regional cerebral oxygen saturation.

DETAILED DESCRIPTION:
The literature includes studies that investigate the relationship of pneumoperitoneum and different positions with intracranial pressure during laparoscopy. Reverse Trendelenburg position has been shown to slightly reduce the intracranial pressure associated with pneumoperitoneum. However, there are no studies on the effect of the timing of reverse Trendelenburg position on intracranial pressure. This study will monitor the effect of reverse Trendelenburg position before or after pneumoperitoneum on intracranial pressure and regional cerebral oxygen saturation. Ultrasound guided measurement of the optic nerve sheath diameter as a non-invasive method will be used for measurement. The investigators believe reverse Trendelenburg position before pneumoperitoneum may prevent undesired sudden increases in intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic cholecystectomy operation
* Age between 18-65
* ASA I-II
* BMI ≤ 35

Exclusion Criteria:

* Ophthalmologic disease and optic nerve pathology
* Increased intracranial pressure
* History of cerebrovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Optic Nerve Sheath Diameter | Throughout the surgery
  The change in intracranial pressure via optic nerve sheath diameter measurement during laparoscopic cholecystectomy among 6 time point.
Change in regional cerebral oxygen saturation | Throughout the surgery
  The change in regional cerebral oxygen saturation during laparoscopic cholecystectomy among 6 time point.

SECONDARY OUTCOMES:
Perioperative Hemodynamic Parameters | Throughout the surgery
  Mean arterial pressure in mmHg
Perioperative Hemodynamic Parameters | Throughout the surgery
  Heart rate beat per minute

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Demirgan, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Robba C, Cardim D, Donnelly J, Bertuccio A, Bacigaluppi S, Bragazzi N, Cabella B, Liu X, Matta B, Lattuada M, Czosnyka M. Effects of pneumoperitoneum and Trendelenburg position on intracranial pressure assessed using different non-invasive methods. Br J Anaesth. 2016 Dec;117(6):783-791. doi: 10.1093/bja/aew356. PMID 27956677
- [Background] Dip F, Nguyen D, Rosales A, Sasson M, Lo Menzo E, Szomstein S, Rosenthal R. Impact of controlled intraabdominal pressure on the optic nerve sheath diameter during laparoscopic procedures. Surg Endosc. 2016 Jan;30(1):44-9. doi: 10.1007/s00464-015-4159-0. Epub 2015 Apr 22. PMID 25899811
- [Background] Sahay N, Sharma S, Bhadani UK, Singh A, Sinha C, Sahay A, Ranjan A, Agarwal M. Effect of Pneumoperitoneum and Patient Positioning on Intracranial Pressures during Laparoscopy: A Prospective Comparative Study. J Minim Invasive Gynecol. 2018 Jan;25(1):147-152. doi: 10.1016/j.jmig.2017.07.031. Epub 2017 Sep 12. PMID 28918894
- [Derived] Demirgan S, Ozcan FG, Gemici EK, Guneyli HC, Yavuz E, Gulcicek OB, Selcan A. Reverse Trendelenburg position applied prior to pneumoperitoneum prevents excessive increase in optic nerve sheath diameter in laparoscopic cholecystectomy: randomized controlled trial. J Clin Monit Comput. 2021 Feb;35(1):89-99. doi: 10.1007/s10877-020-00608-6. Epub 2020 Oct 21. PMID 33089454